CLINICAL TRIAL: NCT00001666
Title: Drug Refractory Partial Epilepsy, A Therapeutic Trial With Transcranial Magnetic Stimulation
Brief Title: Transcranial Magnetic Stimulation for the Treatment of Poorly Controlled Partial Epilepsy
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 970092; 97-N-0092
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2002-06

CONDITIONS: Partial Epilepsy; Seizures
Keywords: Seizures; Partial Epilepsy; Intractable; TMS
MeSH Terms: conditions — Epilepsies, Partial; Seizures

INTERVENTIONS:
Device: Cadwell High-Speed Magnetoelectric Stimulator
Device: Magpro High-Speed Magnetoelectric Stimulator

SUMMARY:
Transcranial Magnetic Stimulation (TMS) is a non-invasive technique that can be used to stimulate brain activity and gather information about brain function. It is very useful when studying the areas of the brain related to motor activity (motor cortex, corticospinal tract, and corpus callosum).

Epilepsy is a condition associated with seizures as a result of an over excitable cerebral cortex. Despite the introduction of several new antiepileptic medications, less than half of the patients diagnosed with partial epilepsy are well controlled. However, studies have shown that non-invasive stimulation of the brain can decrease the excitability of the cerebral cortex.

Researchers are interested in the potential therapeutic effects of TMS on patients with epilepsy that have responded poorly to standard medication. This study will use TMS to decrease the excitability of the areas of the brain responsible for seizures.

DETAILED DESCRIPTION:
The purpose of this protocol is to study the effects of transcranial magnetic stimulation (TMS) at 1 Hz on the excitability of the seizure focus in patients with poorly controlled epilepsy refractory to pharmacological treatments. 1 Hz TMS is a rate proven to induce long term depression in animal models and reported to decrease the excitability of both human and animal cerebral cortex.

ELIGIBILITY:
Age 5 to 60 at entry to protocol.

History of partial or Complex Partial Epilepsy for two or more years.

Patients should be on a stable anti-convulsant regimen defined as unchanged medicines and dose modifications lower than 20% in the last month. Blood levels of anti-convulsants will be measured at the beginning of the study, prior to stimulation and after the study to assure that the type and dose of medication will remain constant.

Seizures not completely responsive to medical treatment (1 or more seizures per week for at least 6 months) and patients have failed at least two anti-convulsant regimens in the past.

The patients have a localized seizure focus.

Epilepsy refractory to medical treatments.

No pregnant women (will be tested with urine pregnancy test).

No severe coronary disease.

No metal anywhere in the cranium except the mouth.

No intracardiac lines.

No increased intracranial pressure as expressed by the presence of papilledema.

No cardiac pacemakers.

Must not be taking neuroleptic or antidepressant medications.

No progressive neurologic disease.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32
Dates: Start 1997-03; Study Completion 2002-06

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States

REFERENCES:
- [Background] Abou-Khalil BW, Siegel GJ, Sackellares JC, Gilman S, Hichwa R, Marshall R. Positron emission tomography studies of cerebral glucose metabolism in chronic partial epilepsy. Ann Neurol. 1987 Oct;22(4):480-6. doi: 10.1002/ana.410220407. PMID 3124709
- [Background] Classen J, Witte OW, Schlaug G, Seitz RJ, Holthausen H, Benecke R. Epileptic seizures triggered directly by focal transcranial magnetic stimulation. Electroencephalogr Clin Neurophysiol. 1995 Jan;94(1):19-25. doi: 10.1016/0013-4694(94)00249-k. PMID 7530636
- [Background] Derby LE, Tennis P, Jick H. Sudden unexplained death among subjects with refractory epilepsy. Epilepsia. 1996 Oct;37(10):931-5. doi: 10.1111/j.1528-1157.1996.tb00529.x. PMID 8822690